CLINICAL TRIAL: NCT00106379
Title: A Phase 4, Single-Arm Study to Evaluate the Safety, Antiviral Activity and Pharmacokinetics of Tenofovir Disoproxil Fumarate in Combination With Emtricitabine in HIV-1 Infected Patients Experiencing Various Degrees of Renal Impairment
Brief Title: Tenofovir DF (Disoproxil Fumarate) in Combination With Emtricitabine in HIV-1 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-104-0235
Record Dates: First submitted 2005-03-23; First posted 2005-03-24 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
Keywords: HIV-1; Treatment Naive; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

INTERVENTIONS:
Drug: Truvada (tenofovir DF + emtricitabine)
Drug: Emtriva (emtricitabine)
Drug: Viread (tenofovir DF)

SUMMARY:
The purpose of this study is to provide long-term clinical safety and efficacy data for tenofovir disoproxil fumarate and emtricitabine in HIV-infected patients experiencing various degrees of renal impairment.

DETAILED DESCRIPTION:
The primary objective of this study is as follows:

* To evaluate the safety and tolerability of tenofovir following administration of tenofovir disoproxil fumarate 300 mg for 48 weeks in HIV-infected patients experiencing various degrees of renal impairment.

The secondary objectives of this study are as follows:

* To evaluate the safety and tolerability of emtricitabine following administration of emtricitabine 200 mg for 48 weeks in HIV-infected patients experiencing various degrees of renal impairment.
* To evaluate the efficacy of tenofovir disoproxil fumarate in combination with emtricitabine in renally-impaired HIV-infected patients.
* To evaluate the pharmacokinetics of tenofovir and emtricitabine in renally-impaired HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in the study.

* HIV-1 infection
* Either antiretroviral therapy-naive requiring antiretroviral treatment with HIV-1 RNA greater than 400 copies/mL or antiretroviral therapy-experienced on a stable antiretroviral regimen for at least 3 mos. with HIV-1 RNA less than or equal to 50 copies/mL at screening.
* No active opportunistic infection within 45 days prior to baseline.
* Able to understand and sign the informed consent form and comply with the study.
* Stable renal impairment within the four defined groups for at least 3 mos., based on creatinine clearance (Cockcroft-Gault method).

Exclusion Criteria:

Patients who meet any of the following are not to be enrolled in this study.

* Women who are pregnant or breastfeeding
* Fanconi syndrome or multiple myeloma, tertiary hyperparathyroidism, malignancy (with the exception of basocellular carcinoma) or myeloproliferative disorder.
* Women of childbearing potential who are unwilling to use an effective contraceptive method during the study
* Contraindications to tenofovir DF, emtricitabine or efavirenz
* Undergoing treatment for tuberculosis
* Using atazanavir
* Prior history of mutation M184V, K65R or T69 insertion
* Z-score on pre-baseline DEXA scan less than -2.5
* The following laboratory values within 30 days prior to study entry: *absolute neutrophil count (ANC) less than 750/mm3, *hemoglobin less than 9.0 g/dL, *platelet count less than 50,000/mm3, *AST (SGOT) or ALT (SGPT) less than 5 x ULN and *CD4 cell count less than 100/mm3.
* Use of nephrotoxic agents or competitors with renal excretions, including aminoglycoside antibiotics, intravenous amphotericin B, cidofovir, cisplatin, foscarnet, intravenous pentamidine, probenecid or other agents with significant nephrotoxic potential
* Clinically significant cardiac, pulmonary or gastrointestinal disorder
* Alcohol or drug abuse that could hinder compliance with the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2004-10; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
HIV-1 infection

SECONDARY OUTCOMES:
HIV-1 infection in renally impaired HIV infected patients

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Gary Richmond, MD, Fort Lauderdale, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Ronald Reisler, MD, Baltimore, Maryland
  - Fernando Garcia, MD, Harlingen, Texas

REFERENCES:
- See also: Truvada website — http://www.truvada.com
- See also: Gilead website — http://www.gilead.com
- See also: Viread website — http://www.viread.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-104-0235_synopsis.pdf